CLINICAL TRIAL: NCT01302951
Title: Study on Pharmacokinetics of Moxifloxacin in Serum and Liver Tissue of Patients Undergoing Liver Resection Due to Primary or Secondary Tumor of the Liver
Brief Title: Penetration of Moxifloxacin Into Liver Tissue of Patients Undergoing Liver Resection.
Acronym: MOXI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Saarland (Other)
Collaborators: Bayer (Industry)
Responsible Party: Martin K Schilling MD, FRCS, University of the Saarland
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 24/06; 2008-001902-18 (EudraCT Number)
Record Dates: First submitted 2011-01-17; First posted 2011-02-24 (Estimated); Last update posted 2011-02-24 (Estimated); Status verified 2011-02

CONDITIONS: Side-effect of Antibiotic
Keywords: pharmacokinetics; liver resection
MeSH Terms: interventions — Moxifloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Moxifloxacin (Experimental): Moxifloxacin 400 mg i.v.
  Interventions: Drug: Moxifloxacin 400 mg
- No drug (No Intervention): 2 Patients were included as controls- no MXF given

INTERVENTIONS:
Drug: Moxifloxacin 400 mg — The patients receive MXF 400 mg as one hour intravenous infusion at randomized timed intervals prior to liver resection.
  Other Names: Avalox 400mg/250ml
  Arms: Moxifloxacin

SUMMARY:
The aim of the study is to provide data on the pharmacokinetics (PK) of moxifloxacin (MXF) in serum and liver tissue of patients undergoing liver resection due to primary or secondary tumor of the liver.

DETAILED DESCRIPTION:
After given informed consent, patients scheduled for planned liver resection are enrolled into the study. The patients receive MXF 400 mg as one hour intravenous infusion at randomized timed intervals prior to liver resection. Blood and healthy liver tissue are sampled in 34 patients after administration of MXF. Plasma is sampled concomitantly. In a subgroup of 19 patients, additional serum specimens are obtained after 2, 4, 8, 12, 24, 36 and 48 h to establish the PK. The pharmacokinetic parameters of MXF are calculated applying a two-compartment model.

ELIGIBILITY:
Inclusion Criteria:

* age 18-80 years old
* elective liver resection of liver tumor
* in females: pregnancy test negative
* Subjects willing and able to give fully informed written consent

Exclusion Criteria:

* subjects with contra-indications to Moxifloxacin
* subjects under therapy with Moxifloxacin within 2 weeks before recruitment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2008-07; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Concentration (mg/L) of moxifloxacin in liver tissue | 1.5 hours after moxifloxacin infusion
  The first outcome of this study was to analyze the concentration of MFX in liver tissue of patients who received MFX 400 mg i.v..

SECONDARY OUTCOMES:
Maximum concentration (mg/L) of moxifloxacin in serum | at the end of intravenous infusion
  The maximum concentration (mg/L) of moxifloxacin in the serum of patients who received 400 mg moxifloxacin was measured at the end of the intravenous infusion.
Number of participants with adverse events | 48 hours
  The number of participants and kind of adverse events were recorded up to 48 hours after intravenous infusion of 400 mg moxifloxacin.
Area under the plasma concentration versus time curve (AUC) of moxifloxacin (mg*h/L) | 48 hours
  The serum concentration of moxifloxacin was measured at different time points (2, 3, 4, 6, 8, 12, 24, 36 hour after infusion) up to 48 hours after intravenous infusion of 400 mg moxifloxacin.

CONTACTS AND LOCATIONS:
Overall Officials: Martin K Schilling, MD, Principal Investigator — University hospital of the Saarland
Locations (1):
- University hospital of the Saarland, Homburg/Saar, Germany

REFERENCES:
- [Background] Weinrich M, Scheingraber S, Stremovskaia T, Schilling MK, Kees F, Pistorius GA. Liver tissue concentrations of levofloxacin after single intravenous administration of 500 mg for antibiotic prophylaxis in liver surgery. Int J Antimicrob Agents. 2006 Sep;28(3):221-5. doi: 10.1016/j.ijantimicag.2006.04.012. Epub 2006 Aug 14. PMID 16904875
- [Derived] Justinger C, Schilling MK, Kees MG, Kauffels A, Hirschmann K, Kopp B, Kees F, Kollmar O. Penetration of moxifloxacin into liver tissue. Int J Antimicrob Agents. 2012 Jun;39(6):505-9. doi: 10.1016/j.ijantimicag.2012.01.022. Epub 2012 Apr 21. PMID 22526014
- See also: PI´s institute homepage — http://www.uniklinikum-saarland.de/de/einrichtungen/kliniken_institute/chirurgie/allgemeinchirurgie/